CLINICAL TRIAL: NCT06750016
Title: Non-invasive Detection of Coronary Artery Stenosis
Acronym: NIDCAS
Status: Not yet recruiting | Type: Observational
Sponsor: Nilocas (Industry)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Stephen Greenwald, Professor of Cardiovascular Mechanics, Nilocas
Other Study IDs: NIDCAS002
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Stenosis; Turbulent flow; Acoustic signature
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease (CAD): Patients in whom occlusive coronary artery disease has been diagnosed by angiography or CT angiography
- Control: Healthy volunteers and/or patients in whom no CAD has been identified on angiography or CT angiography

SUMMARY:
The aim of this viability study is to investigate using a novel medical device, the potential for detecting partial blockages in the arteries within the wall of the heart (coronary artery stenosis). A prototype device will be used in the proposed study. It is a stick-on patch containing sensors which measure the vibration produced at the chest surface by flowing blood as it accelerates through the narrowed artery in the heart emerging downstream, hitting the inner wall of the artery and causing it to vibrate. Some of the energy in the vibrations reaches the skin of the chest, allowing the blockage to be detected non-invasively. The principle has been proved in the laboratory using a simple chest model but to date no measurements have been made in people. Therefore, the proposed trial will serve as the first in-human measurements and will involve a small number of patients and healthy volunteers, with the objective of establishing if it is possible to determine the presence or absence of the stenosis.

The patch will be tested by recording acoustic signatures in healthy volunteers, then in patients undergoing coronary CT angiography. Results will be validated against the CT angiography gold standard. At this early stage no clinical decisions will be made based on the patch recordings and the data will be used only to assess the feasibility of continuing the development of the device.

DETAILED DESCRIPTION:
This feasibility study is a non-randomised, proof of concept study being undertaken at a single clinical centre. It involves a novel, non-invasive battery powered medical device that is not CE marked. As a non-CE marked device, review and approval of the proposed clinical investigation a UK Competent Authority, the HRA, is required in addition to ethical review and approval.

The device, a patch containing microphones and accelerometers applied to the chest, is battery powered and will not introduce any energy or substances into the subjects involved in the study. The device will listen for sounds and movement within the body of the individual being examined. The signals detected by the microphones and accelerometers are transmitted wirelessly to a data acquisition unit which is connected to a laptop computer more than 2 metres away from the patient, which displays the signals in real time and stores them for later analysis off-line.

Data (acoustic signatures) will be collected from patients with known or suspected coronary artery disease. Results will be compared with the current gold standard of coronary angiography or coronary CT angiography.

The risk to participants is minimal. No specific risks associated with the use of the device have been identified and no requirement for additional testing has been identified. There are no anticipated interactions with concomitant medical treatments.

The results of this study will not be used to manage the treatment pathway of the patient involved.

If proof of concept is successfully demonstrated with the new device, a larger randomised study will be undertaken to obtain the clinical data necessary to support commercial and regulatory requirements.

Having conducted in-vitro proof of principle experiments (as listed in the references section) and before conducting a formal validation trial, we wish to determine the viability of the new patch device in an initial study on a small number of patients undergoing coronary angiography. We aim firstly, to prove the principle that it is possible to distinguish between those with and those without coronary artery stenosis and, secondly to assess how well the device is tolerated by the patient and how easy it is to deploy the patch and take readings 'in the field'. We believe that this small trial is essential to provide first in human data to support applications for funding a larger validation trial.

Potential study participants will be recruited from patients attending, the Cleveland Clinic who have agreed to elective angiography or CTa investigation. All potential participants will be screened against the inclusion and exclusion criteria detailed elsewhere. This is a non-randomised study. Accordingly, participants will be recruited i on a sequential basis until a total sample size of at least 20 is reached.

Written Informed Consent will be obtained from all participants before recruitment into the study and this will be recorded on the consent form. The nature of the measurements and the nature of the clinical investigation, together with all procedures and risks will be fully explained to each prospective participant by one of the Investigators or members of the research team. If the patient meets all inclusion/exclusion criteria and agrees to participate in the study, he/she will be invited to sign the approved CF.

When the potential subject has agreed to take part, they will undergo the following procedures (approximate times in brackets).

* Height, weight and blood pressure recording. (15 minutes)
* CTa or angiography scan as normal. (30 minutes)
* Patch attached and wireless connection to remote receiver established.
* The patch will be adjusted to ensure that the patient is comfortable
* Data recorded. (15 minutes)
* Patch removed. (5 minutes)
* Subject asked to suggest any aspects of the procedure that might be improved. All comments noted. (10 minutes)

The patch data will be analysed blind by a member of our team who would not take part in the recording sessions. For the analysis the time series data will be transformed to the frequency domain and the relative acoustic power detected by each sensor over various frequency range will be tabulated. For this small preliminary study, the agreement between the reference and test method to determine the categorical variable namely, the presence or absence of a coronary artery stenosis, will be assessed by Cohen's Kappa test. This measures how much the agreement between the two methods exceeds what would be expected by chance. At this early stage no further statistical tests are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written informed consent
2. Age ≥18 years;
3. Investigation for suspected stable coronary artery disease/stenosis isolated from other cardiac comorbidities.
4. Subjects of either sex. Female subjects of child-bearing potential will be included if deemed suitable for clinically mandated coronary CTa.
5. No infectious disease or neoplasia.

Exclusion Criteria:

1. Indications to coronary CTa different from isolated suspected stable coronary artery disease, such as acute coronary syndrome, unstable angina, congenital heart disease, cardiomyopathy, heart valve disease, aortic coarctation, electrophysiological disorder/arrhythmia, screening study, unstable clinical condition, left ventricular ejection fraction <35%, previous coronary revascularization (PCI or CABG surgery), previous heart valve surgery or transcatheter valve replacement, pace maker or implantable defibrillator.
2. If female and of child-bearing potential: evidence of a positive pregnancy test or a stated intention to become pregnant in the next 6-12 months;
3. Currently participating in another device or drug study or has done so in previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately equal numbers of symptomatic and asymptomatic subjects undergoing angiography or CT angiography at the Cleveland Clinic, London, UK
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Immediately following patch recording and imaging
  Diagnostic accuracy of the device (stick-on patch) for indicating the presence or absence of one or more coronary arterial stenoses as indicated by the reference method (angiography/CT angiography results). This will be expressed as: Np/(Na+Np) x100.
  Where:
  Np is the number of positive diagnoses of coronary artery disease derived from the patch measurements Na is the number of positive diagnoses of coronary artery disease (with at least one lesion showing a reduction in maximum stenosis lumen diameter 0.8 of more) derived from the angiography images.
  This is a dimensionless quantity

SECONDARY OUTCOMES:
Stenosis severity | Immediately following the patch recordings and imaging
  In subjects in whom one or more stenoses are identified by the reference method:
  Comparison of the magnitude of the disturbed flow to the severity of the stenosis as measured from the CTa images.
  The comparison will be made by assessing the significance of the linear correlation coefficient between the average power of the patch signals in the frequency domain (in the frequency range 20 - 500 Hz) and the stenosis severity defined as the ratio of the minimum stenosis diameter to the mean diameter of the coronary artery immediately proximal to the stenosis. (Note that this is at best, a semi-quantitative measure and with the small number of subjects proposed for this viability trial the results are for guidance only.)
Patch wearability | Immediately following the patch recordings and imaging
  Assessment of the subject's comfort when wearing the device. This will be quantified using a Visual Analog Score between 1 and 10, 1 being the least comfortable and 10, the most.
Ease of patch removal | Immediately following the patch recordings and imaging
  Ease of removal at the end of a measurements session. This will be quantified quantified using a Visual Analog Score between 1 and 10, 1 being the least comfortable and 10, the most.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Pugliese, MD, Principal Investigator — Queen Mary University of London
Locations (1):
- Cleveland Clinic Portland Place Outpatient Centre 24 Portland Place, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results of this preliminary viability study will be described in an internal report and this will be used to provided evidence when seeking funding for a larger validation trial. They will not therefore be published.

REFERENCES:
- [Background] Banks HT, Hu S, Kenz ZR, Kruse C, Shaw S, Whiteman J, Brewin MP, Greenwald SE, Birch MJ. Model validation for a noninvasive arterial stenosis detection problem. Math Biosci Eng. 2014 Jun;11(3):427-48. doi: 10.3934/mbe.2014.11.427. PMID 24506547
- [Background] Brewin MP, Birch MJ, Mehta DJ, Reeves JW, Shaw S, Kruse C, Whiteman JR, Hu S, Kenz ZR, Banks HT, Greenwald SE. Characterisation of Elastic and Acoustic Properties of an Agar-Based Tissue Mimicking Material. Ann Biomed Eng. 2015 Oct;43(10):2587-96. doi: 10.1007/s10439-015-1294-7. Epub 2015 Mar 14. PMID 25773982
- [Background] Sangster JF, Oakley CM. Diastolic murmur of coronary artery stenosis. Br Heart J. 1973 Aug;35(8):840-4. doi: 10.1136/hrt.35.8.840. No abstract available. PMID 4542336
- [Background] Semmlow J, Rahalkar K. Acoustic detection of coronary artery disease. Annu Rev Biomed Eng. 2007;9:449-69. doi: 10.1146/annurev.bioeng.9.060906.151840. PMID 17425468